CLINICAL TRIAL: NCT06350929
Title: Evaluation of Norepinephrine in the Management of General Anesthesia-Induced Arterial Hypotension in Chronic Heart Failure Patients in the Operating Room.
Brief Title: Norepinephrine in the Management of General Anesthesia-Induced Arterial Hypotension in Chronic Heart Failure Patients
Acronym: NORAFLOW
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0017
Record Dates: First submitted 2024-03-28; First posted 2024-04-08 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Hypotension
Keywords: Chronic heart failure; Norepinephrine; General anaesthesia
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Research procedures: Patients with heart failure
  Interventions: Other: Cardiac output monitoring by the Starling™ SV Sebac®

INTERVENTIONS:
Other: Cardiac output monitoring by the Starling™ SV Sebac® — During the surgery, the channels and monitoring equipment will be set up according to the usual procedure in the vascular surgery department. As part of the research, the Starling™ SV Sebac® electrodes will be installed (to measure cardiac flow, cardiac index (CI), stroke volume (VES), variations in stroke volume (VVES), and peripheral resistors (TPRI)).
  Once the equipment is in place, anesthetic induction will be carried out according to the usual protocol with curarization and mechanical ventilation.
  If the appearance of arterial hypotension is noted after anesthetic induction and mechanical ventilation, the patient will be definitively included in the study. As recommended, he will receive norepinephrine to treat hypotension.
  The measurements from the monitoring will be collected at 3, 5, and 10 min after the administration of norepinephrine.
  10 days after admission to the operating room, hospitalization data will be collected.

SUMMARY:
Arterial hypotension is a frequent complication of general anesthesia and a significant contributor to postoperative complications. It is a critical marker for the development of acute renal failure and postoperative myocardial infarction. Chronic heart failure (CHF) patients are increasingly encountered in the operating room, and their perioperative morbidity and mortality are substantial, with specific management lacking precise recommendations.

The main objective is to assess the impact of a diluted norepinephrine bolus on cardiac output in chronic heart failure patients experiencing arterial hypotension after anesthesia induction.

DETAILED DESCRIPTION:
Arterial hypotension is a frequent complication of general anesthesia and a significant contributor to postoperative complications. It is a critical marker for the development of acute renal failure and postoperative myocardial infarction. Chronic heart failure (CHF) patients are increasingly encountered in the operating room, and their perioperative morbidity and mortality are substantial, with specific management lacking precise recommendations. The potential indications for norepinephrine use are expanding due to dilution methods allowing peripheral catheter administration, particularly for addressing arterial hypotension during general anesthesia induction. However, these indications are primarily based on common practices, and the impact of norepinephrine on cardiac output in patients with chronic heart failure is poorly understood. The main objective is to assess the impact of a diluted norepinephrine bolus on cardiac output in chronic heart failure patients experiencing arterial hypotension after anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Heart failure patients with left ventricular failure with a ventricular ejection fraction less than or equal to 40% evaluated by trans-thoracic echocardiography less than a year ago and specifying in particular the patient's filling pressures at the state stable.
* Patients under treatment adapted to the level of heart failure according to the 2021 European Society of Cardiology recommendations.
* Scheduled surgery under general anesthesia.
* Invasive hemodynamic monitoring planned by the anesthetist-resuscitator (irrespective of potential inclusion in the protocol): arterial catheter and central venous line for measurement of CVP (central venous pressure).
* Postoperative monitoring planned in intensive care or intensive care
* Presence of controlled mechanical ventilation with tidal volumes between 8 and 10 ml/kg of ideal weight.
* Presence of arterial hypotension after induction of general anesthesia, and before surgical stimulation.
* Patient affiliated to a social security scheme or equivalent
* No opposition from the patient.

Exclusion Criteria:

* Chronic heart failure patients with right ventricular failure.
* Patients presenting signs of acute pulmonary edema, Pulmonary arterial hypertension (PAH), severe valvular disease, intracardiac shunt.
* Patients operated on under general anesthesia but maintaining spontaneous ventilation.
* Patients with respiratory compliance disorders with compliances greater than 30 cm of water.
* Patients with intra-abdominal hypertension.
* Patients with supraventricular or ventricular arrhythmia.
* Patients treated with catecholamines prior to the procedure.
* Patients operated on for urgent surgeries
* Patient under guardianship, curatorship or safeguard of justice
* Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with heart failure and left ventricular failure with a ventricular ejection fraction less than or equal to 40%.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the impact of a bolus of diluted norepinephrine on cardiac output in chronic heart failure patients presenting with arterial hypotension after anesthetic induction. | During the surgery.
  The evolution of the value of cardiac output assessed by non-invasive monitoring, using bioreactance: Starling™ SV Sebac®.

SECONDARY OUTCOMES:
Evaluation of the role of preload dependence before anesthetic induction in the variation of cardiac output after a norepinephrine bolus. | During the surgery.
  Measurement of pulse pressure difference.
Evaluation of the impact of the norepinephrine bolus on blood pressure correction. | During the surgery.
  Evolution of the monitoring data: systolic blood pressure (SBP - mmHg).
Evaluation of the impact of the norepinephrine bolus on heart rate. | During the surgery.
  Evolution of the monitoring data: heart rate (HR - bpm).
Evaluation of the safety of use of norepinephrine in chronic heart failure patients during hospitalization. | For 10 days after surgery.
  Monitoring the appearance of side effects during post-operative hospitalization on the assessments usually carried out in the department and including.

CONTACTS AND LOCATIONS:
Overall Officials: François LABASTE, Dr, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse Rangueil, Toulouse, France

IPD SHARING:
Plan to Share IPD: No